CLINICAL TRIAL: NCT04291885
Title: A Randomised, Placebo-controlled, Phase II Trial of Adjuvant Avelumab in Patients With Stage I-III Merkel Cell Carcinoma
Brief Title: Immunotherapy Adjuvant Trial in Patients With Stage I-III Merkel Cell Carcinoma
Acronym: I-MAT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Melanoma and Skin Cancer Trials Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03.18
Record Dates: First submitted 2020-02-06; First posted 2020-03-02 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Merkel Cell Carcinoma; Merkel Cell Carcinoma, Stage I; Merkel Cell Carcinoma, Stage II; Merkel Cell Carcinoma, Stage III; Neuroendocrine Tumors; Carcinoma Neuroendocrine Skin
MeSH Terms: conditions — Carcinoma, Merkel Cell; Neuroendocrine Tumors | interventions — avelumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Avelumab (Experimental): 6 months of Avelumab at a dose of 800mg as a 60-minute intravenous (IV) infusion once every 2 weeks (13 doses)
  Interventions: Drug: Avelumab
- Placebo (Placebo Comparator): 6 months of Placebo as a 60-minute intravenous (IV) infusion once every 2 weeks (13 doses)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avelumab — Avelumab IV infusion
  Other Names: anti-PD-L1; Bavencio
  Arms: Avelumab
Drug: Placebo — Placebo IV infusion
  Arms: Placebo

SUMMARY:
The I-MAT trial is a randomised, placebo-controlled, phase II trial of adjuvant Avelumab in patients with stage I-III Merkel cell carcinoma aiming to explore the efficacy of avelumab as adjuvant immunotherapy.

DETAILED DESCRIPTION:
The I-MAT trial is a phase II, prospective, randomised, placebo-controlled, multi-institutional trial for patients with stage I-III Merkel cell carcinoma (MCC). Participants on the trial will receive either avelumab or placebo for 6 months. The primary aim of the I-MAT trial is to develop an effective, well-tolerated adjuvant immunotherapy regimen for patients with stage I-III MCC, post a range of definitive loco-regional treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Merkel cell carcinoma (MCC) which is either:

   * clinical stage I;
   * pathological stage I with positive LVSI only;
   * clinical or pathological stage II (including IIA and IIB);
   * clinical or pathological stage III (including IIIA and IIIB).
2. Absence of distant metastatic disease on baseline 18-Fludeoxyglucose (18FDG) - Positron Emission Tomography (PET) / Computed Tomography (CT) scan.
3. 18 years of age or older.
4. Eastern Cooperative Oncology Group (ECOG) of 0 - 2.
5. Willing and able to provide written informed consent and comply with all study requirements.
6. Adequate haematological, liver and renal function as determined by the screening laboratory values outlined in the protocol obtained within 14 days prior to randomisation.
7. Agreeable to collection of archival tumour material. Where possible, the most recently acquired tumour specimen should be provided.
8. Women of child bearing potential (WOCBP) must have a negative serum or urine pregnancy test within 72 hours prior to the start of treatment.

Exclusion Criteria:

1. Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest significant risk for immune-related adverse events.
2. Prior treatment with an agent that blocks the PD-1/PD-L1 pathway.
3. Previous cancer immunotherapy, specifically interferon, anti-CD137, or anti-CTLA-4 antibody or any other antibody or drug specifically targeting T cell co-stimulation or checkpoint pathways are not permitted.
4. Prior treatment with other immune-modulating agents that was within fewer than 28 days prior to the first dose of Avelumab.
5. Active infection requiring antibiotics within 7 days of cycle 1 day 1 of study drug dose.
6. Active tuberculosis.
7. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
8. Uncontrolled infection with hepatitis B or hepatitis C virus (HBV or HCV) infection; Patients with previously successfully treated HCV, with positive anti-HCV antibody but undetectable (HCV) ribonucleic acid (RNA) levels are allowed on trial.
9. Current use of immunosuppressive medication, except for the following: a. intranasal, inhaled, topical steroids, or local steroid injection ; b. systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. steroids as premedication for hypersensitivity reactions
10. Any systemic anti-cancer treatment (chemotherapy, targeted systemic therapy) investigational or standard of care, within 28 days of the first dose of Avelumab or planned to occur during the study period. Patients receiving bisphosphonates or denosumab will not be excluded.
11. Pregnant or breastfeeding.
12. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organising pneumonia (i.e., bronchiolitis obliterans, cryptogenic organising pneumonia), or evidence of active pneumonitis on screening chest CT scan).
13. Uncontrolled cardiac disease including not limited to symptomatic congestive heart failure, unstable angina pectoris, life-threatening cardiac arrhythmia
14. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5 Grade 3).
15. Use of live attenuated vaccines within 28 days of first dose of Avelumab.
16. Any acute or chronic psychiatric problems that, in the opinion of the Investigator, make the patient ineligible for participation due to compliance concerns.
17. Patients with prior allogeneic stem cell or solid organ transplantation.
18. Patients who are involuntarily incarcerated.
19. Evidence of other malignancy in the past 3 years, with exception of tumours with negligible risk of metastasis or death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | 24 Months
  Recurrence-free survival (RFS) as the primary endpoint, is anticipated to be analysed over an average planned follow-up of 3.5 years. An analysis of RFS at the 24 month time point of follow-up will also be conducted as it is anticipated that the minimum follow-up for participants will be 24 months and the sample size rationale utilises RFS rates at 24 months in historical controls. RFS is defined as the time from treatment initiation until the first date of any signs or symptoms of recurrence of tumour.

SECONDARY OUTCOMES:
Overall survival (OS) | 24 Months
  Overall survival rates at 12 and 24 months. Overall survival is defined as the time from treatment initiation to the date of death due to any cause.
Disease-specific survival (DSS) | 24 Months
  Disease-specific survival at 24 months from treatment initiation. Disease-specific survival is the percentage of participants who have not died from Merkel Cell Carcinoma
Rate of loco-regional failure free survival (LRFFS) | 24 Months
  Rate of loco-regional failure free survival (LRFFS) is defined as the time from treatment initiation to the first recurrence of the loco-regional tumour.
Distant metastasis-free survival (DMFS) | 24 Months
  DMFS is defined as the time from treatment initiation to the first evidence of distant metastatic disease.
Treatment toxicity and tolerability as assessed by NCI CTCAE v5.0 | 24 Months
  Rate of treatment-related adverse events (AEs). Safety will be measured by serious adverse events (SAEs) and AEs assessed as per NCI CTCAE v5.0, including immune-related adverse events.
Patient-reported quality of life (QoL) as assessed by FACT-M questionnaire | 24 Months
  FACT-M form (version 4) will be utilised. This will include patient-reported questions relating to physical wellbeing, social/family wellbeing, emotional wellbeing, functional wellbeing and additional patient concerns which are measured from 0-4 (Not at all - Very Much).

OTHER OUTCOMES:
Rate of Merkel cell polyomavirus positivity in stage I-III Merkel cell carcinoma | 24 Months
  To identify Merkel cell polyomavirus MCPyV virus status. To correlate viral aetiology-rate of Merkel cell polyomavirus (MCPyV) positivity in pathology specimens in stage I-III Merkel cell carcinoma with outcome from adjuvant treatment.
Correlating whole exome sequencing (WES) and ribonucleic acid (RNA) expression with immunotherapy response and outcomes in early stage MCC | 24 Months
  To evaluate the relationship between somatic mutations in cancer genes or the total mutation burden of the cancer with immunotherapy response and outcome following adjuvant therapy.
Correlating immune infiltrates by multiplex immunohistochemistry (IHC) with survival endpoints | 24 Months
  To address whether immune infiltrates and PD-L1 expression are associated with survival.
Utility of circulating biomarkers in predicting recurrence in early stage MCC | 24 Months
  To identify predictive biomarkers for response and resistance to immunotherapy in patients with stage I-III MCC using archival tissue and peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof Wen Xu, MBBS, FRACP, Study Chair — Princess Alexandra Hospital
Locations (20):
- Australia (19):
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Chris O'Brien Lifehouse, Sydney, New South Wales
  - Melanoma Institute Australia, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Calvary Mater Hospital, Sydney, New South Wales
  - Cancer Care Wollongong, Wollongong, New South Wales
  - Royal Brisbane and Woman's Hospital, Brisbane, Queensland
  - Cancer Care Service, Bundaberg Base Hospital, Bundaberg, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Cancer Care Service, Hervey Bay Hospital, Hervey Bay, Queensland
  - Mackay Hospital and Health Service, Mackay, Queensland
  - Tasman Health Care, Southport, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Icon Cancer Centre Hobart, Hobart, Tasmania
  - Alfred Hospital, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No